CLINICAL TRIAL: NCT05609253
Title: Itraconazole Repurposing to Reduce Residual Cancer Risk in Patients With High-risk Barrett's Esophagus After Ablation
Brief Title: Itraconazole to Prevent Recurrent Barrett's Esophagus
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Texas, Southwestern Medical Center at Dallas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00148341
Record Dates: First submitted 2022-09-26; First posted 2022-11-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Barrett Oesophagitis With Dysplasia
Keywords: Barrett's esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: The primary purpose is to determine the ideal formulation (capsule versus solution) of itraconazole in this short-term pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Itraconazole in capsule form (Active Comparator): Participants in this arm will receive the capsule form of itraconazole
  Interventions: Drug: Itraconazole in capsule form
- Itraconazole in solution form (Active Comparator): Participants in this arm will receive the solution form of itraconazole
  Interventions: Drug: Itraconazole in solution form

INTERVENTIONS:
Drug: Itraconazole in capsule form — Patients with high-risk BE will receive two weeks of itraconazole in the capsule form (N=5).
  Arms: Itraconazole in capsule form
Drug: Itraconazole in solution form — Patients with high-risk BE will receive two weeks of itraconazole in the solution form (N=5).
  Arms: Itraconazole in solution form

SUMMARY:
Recurrent Barrett's esophagus (BE) that occurs at the rate of 12.4%/year is the Achilles heel of the endoscopic treatment of high-risk BE. Over time, after eradication, BE ultimately recurs in as many as 30-50% of the patients putting them at risk for esophageal adenocarcinoma (EAC), thereby undoing the benefits of an effective initial therapy. Also, recurrences need retreatments that increase costs and complications including strictures and refractory ulcerations. A therapy to prevent recurrent BE does not currently exist. Itraconazole with its ability to inhibit important molecular pathways related to BE development could enhance the long-term effectiveness of endoscopic eradication of high-risk BE, thereby promoting a long-term cure

ELIGIBILITY:
Inclusion Criteria:

* Patients with Barrett's esophagus with either confirmed low-grade dysplasia or high grade dysplasia or intramucosal/T1 adenocarcinoma (see histologic review) being considered for endoscopic treatment. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

* Inability to provide informed consent, New York Heart Association class III or IV congestive heart failure (CHF), liver function tests (LFT)>3X upper limit of normal, drug allergy to itraconazole, pregnancy, prolonged QTc (>450 ms for men and QTc>470 ms for women) or critical drug interactions with other medications metabolized by cytochrome P450(CYP)3A4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Itraconazole drug and blood levels | 8-12 months after study initiation
  The primary endpoint will be the tissue (in esophageal biopsies) and blood concentrations of itraconazole.

SECONDARY OUTCOMES:
Safety and tolerability of itraconazole | 8-12 months after study initiation
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Effects of itraconazole on Gli1 expression | 8-12 months after study initiation
  Reduction in Gli1 expression
Effects of itraconazole on (Patched) PTCH expression | 8-12 months after study initiation
  Reduction in PTCH expression by IHC
Effects of itraconazole on AKT pathway | 8-12 months after study initiation
  Reduction in Phospho S6 by IHC
Effects of itraconazole on angiogenesis | 8-12 months after study initiation
  Reduction in Vascular endothelial growth factor (VEGF)/ Vascular endothelial growth factor receptor type 2 (VEGFR2) by IHC

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided